CLINICAL TRIAL: NCT07146529
Title: Study of the Prevalence of Transmitted HIV-1 Resistance, Viral Diversity, and Cluster Identification in Patients at the Time of HIV-1 Diagnosis
Acronym: PRINAVIH
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: INSERM UMR S 1136 (Other); iPLesp (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS0789s PRINAVIH
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HIV Seropositivity; HIV Drug Resistance; HIV Infections
Keywords: Genotyping; HIV-1; HIV drug resistance; Transmitted resistance; Viral diversity; Transmission clusters; Primary infection
MeSH Terms: conditions — HIV Seropositivity; HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to determine the frequency of transmission of viruses carrying at least one antiretroviral resistance mutation in all participants newly diagnosed with HIV-1

DETAILED DESCRIPTION:
This is a national, multicenter, cross-sectional study with both retrospective and prospective data collection :

Retrospective phase (2019-2024): Data will be collected from all participants diagnosed at the time of primary HIV-1 infection during these six years.

Prospective phase (2025-2035): Data will be collected from all participants newly diagnosed with HIV-1, regardless of whether they are at the stage of primary infection.

The study will be offered to all virology laboratories that participated in the last quality control of genotyping of the resistance group of the ANRS MIE virology laboratory network.

For ten years, the virology laboratories that participated in the last quality control of HIV resistance genotyping of the ANRS MIE Virology network will be asked to systematically include all patients meeting the inclusion criteria. The virology laboratories must send the list of eligible patients to the associated clinical centers, according to their usual data transfer procedure, so that they can inform the participants and obtain their consent. An information form will then be distributed to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) aged 18 years or older ;
* Participant newly diagnosed in the laboratory, for whom mandatory HIV seropositivity reporting to Santé Publique France (SPF) is required ;
* Participant naïve to all antiretroviral treatments (except PrEP and/or post-exposure prophylaxis [PEP]) ;
* Participant with an available HIV resistance genotype, including amplification of at least reverse transcriptase and protease ;
* Participant who has not objected to participating in the study.

Exclusion Criteria:

* Participant who objects to the use of their data ;
* Participant currently on antiretroviral treatment ;
* Participant subject to legal protection measures (safeguard of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult participants (male or female) aged 18 years or older, newly diagnosed with HIV-1 in participating laboratories where mandatory reporting to Santé Publique France (SPF) is required. Participants must be antiretroviral treatment-naïve (except for PrEP or PEP) and have an available HIV resistance genotype including amplification of at least reverse transcriptase and protease. Participants who have not objected to participation in the study are eligible. Excluded are participants currently on antiretroviral treatment, those who object to the use of their data, and individuals under legal protection measures (safeguard of justice)
Sampling Method: Probability Sample
Enrollment: 30060 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2036-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment-naïve or acutely infected participants with a virus carrying at least one antiretroviral resistance mutation | At baseline (at the time of HIV diagnosis)
  Data will be collected once, at the time of HIV diagnosis. The participant's genotypic resistance test is performed locally and is part of the standard pre-therapeutic assessment.
  The presence of resistance mutations will be defined by the identification of at least one resistance mutation included in the Stanford and IAS resistance mutation lists. Antiretroviral resistance will be analyzed using the latest versions of the ANRS and Stanford algorithms.
  The χ² (chi-square) or Fisher exact test will be used to compare categorical variables and the Mann Whitney test will be used to compare continuous variables between groups. 95% confidence intervals will be constructed for each calculated proportion. Univariate and multivariate logistic regression models will be used to identify the factors associated with the detection of viruses resistant or possibly resistant to antiretrovirals. The statistical tests will be bilateral with a significance threshold set at 5%.

IPD SHARING:
Plan to Share IPD: No